CLINICAL TRIAL: NCT00917085
Title: Self-Regulatory Preterm Infant Care: Adaptation Postbirth
Brief Title: Is Skin-to-Skin Care Helpful for Preterm Infants and Their Mothers After Birth?
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Gene Cranston Anderson, PhD, RN, FAAN, Case Western Reserve University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2R01NR002444-04A1 (NIH); M01RR000080 (NIH)
Record Dates: First submitted 2009-06-08; First posted 2009-06-10 (Estimated); Last update posted 2009-08-10 (Estimated); Status verified 2009-08

CONDITIONS: Moderate to Late Prematurity
Keywords: Preterm infant; Skin-to-skin contact; kangaroo care; temperature; behavioral state
MeSH Terms: conditions — Premature Birth | interventions — Kangaroo-Mother Care Method

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (No Intervention): Control infants received the same standard care as infants who were not in the study. Infants were kept warm in incubators or warmer beds and were wrapped in blankets when held by their mothers. Hospital staff was responsible for providing standard care.
- Skin-to-Skin group (Experimental)
  Interventions: Behavioral: Skin-to-Skin contact

INTERVENTIONS:
Behavioral: Skin-to-Skin contact — Infants in the Skin-to-Skin group also had standard care provided by hospital staff. In addition, the researchers facilitated skin-to-skin contact by placing diaper-clad infants prone between their mothers' breasts as soon as possible after birth. Thereafter the infants and their mothers experienced skin-to-skin contact as often as possible and for as long as possible each time throughout the protocol.
  Other Names: Kangaroo Care
  Arms: Skin-to-Skin group

SUMMARY:
To see if infant outcomes will improve when mothers are helped to hold their preterm infants skin-to-skin as soon as possible after birth and as often as possible and for as long as possible each time during the next five days.

DETAILED DESCRIPTION:
A similar intervention was studied in a RCT with fullterm infants but this was done with emphasis on close contact rather than skin-to-skin contact and lasted only the first 6 hours postbirth. This study was conducted by the same PI and funded by the National Center for Nursing Research, NIH 1990-1994. This research yielded numerous significant and beneficial differences.

Two pilot studies were done with healthy late preterm infants and mothers who planned to breastfeed. Skin-to-skin contact began in the delivery room. The first pilot was a descriptive exploratory study with 10 mother-infant dyads done in Cali, Colombia; skin-to-skin began at birth and lasted through hour 6 when all dyads went to the postpartum ward. Follow-up was through hospital discharge on the second day. All outcomes were positive.

The second pilot was an RCT done in the United States with a well balanced sample of 8 dyads, 4 in each group. Mean observation time lasted 47 hours (Medicaid required discharge time for the mothers) with skin-to-skin contact occurring 84% of the time. All outcomes favored the skin-to-skin group, for example 3.8 days to discharge home compared to 14.5 for the controls. Follow-up was at one year and similarly positive.

Similar differences were hypothesized for the RCT reported here in which the intervention was extended to the care of somewhat smaller and sicker preterm infants and lasted five days unless the infant was discharged sooner. The consent form was in layman terms, four pages long, and fulfilled all the requirements of the Institutional Review Boards of the Bolton School of Nursing at Case Western Reserve University, University Hospitals Case Medical Center and its General Clinical Research Center, and Kadlec Medical Center, Richmond, WA.

ELIGIBILITY:
Inclusion Criteria:

Mother and Infant Dyads

Infants:

* singleton birth
* 32 to 36 completed weeks
* 5-minute Apgar score of 6 or more
* weighed 1300 to 3000 grams
* no birth defects that would interfere with feeding
* healthy enough to experience skin-to-skin contact with their mothers.

Mothers:

* 18 or more years of age
* spoke English
* free of serious drug abuse
* well enough to experience skin-to-skin contact with their infants with assistance if needed.

Exclusion Criteria:

Infants:

* too ill to be with their mothers
* who have a condition that interferes with feeding.

Mothers:

* who are too ill to care for their infant
* are serious drug abusers.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 1996-07; Primary Completion 2001-12 (Actual); Study Completion 2001-12 (Actual)

PRIMARY OUTCOMES:
Infant Temperature | A total of 60 measrements for each outcome beginning at birth once every 15 minutes and gradually decreasing in frequency to once every 6 hours by Day 5.

SECONDARY OUTCOMES:
Infant Behavioral State | A total of 60 measrements for each outcome beginning at birth once every 15 minutes and gradually decreasing in frequency to once every 6 hours by Day 5.

CONTACTS AND LOCATIONS:
Overall Officials: Gene C Anderson, PhD, RN, FAAN, Principal Investigator — Case Western Reserve University
Locations (2):
- United States (2):
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - Kadlec Medical Center, Richmond, Washington

REFERENCES:
- [Background] Moran M, Radzyminski SG, Higgins KR, Dowling DA, Miller MJ, Anderson GC. Maternal kangaroo (skin-to-skin) care in the NICU beginning 4 hours postbirth. MCN Am J Matern Child Nurs. 1999 Mar-Apr;24(2):74-9. doi: 10.1097/00005721-199903000-00006. PMID 10083783
- [Background] Anderson GC, Dombrowski MA, Swinth JY. Kangaroo care: not just for stable preemies anymore. Reflect Nurs Leadersh. 2001;27(2):32-4, 45. No abstract available. PMID 11987376
- [Background] Dombrowski MA, Anderson GC, Santori C, Burkhammer M. Kangaroo (skin-to-skin) care with a postpartum woman who felt depressed. MCN Am J Matern Child Nurs. 2001 Jul-Aug;26(4):214-6. doi: 10.1097/00005721-200107000-00012. PMID 11452667
- [Background] Anderson GC, Chiu SH, Dombrowski MA, Swinth JY, Albert JM, Wada N. Mother-newborn contact in a randomized trial of kangaroo (skin-to-skin) care. J Obstet Gynecol Neonatal Nurs. 2003 Sep-Oct;32(5):604-11. doi: 10.1177/0884217503256616. PMID 14565739
- [Background] Swinth JY, Anderson GC, Hadeed AJ. Kangaroo (skin-to-skin) care with a preterm infant before, during, and after mechanical ventilation. Neonatal Netw. 2003 Nov-Dec;22(6):33-8. doi: 10.1891/0730-0832.22.6.33. PMID 14700180
- [Background] Hake-Brooks SJ, Anderson GC. Kangaroo care and breastfeeding of mother-preterm infant dyads 0-18 months: a randomized, controlled trial. Neonatal Netw. 2008 May-Jun;27(3):151-9. doi: 10.1891/0730-0832.27.3.151. PMID 18557262
- [Background] Chiu SH, Anderson GC. Effect of early skin-to-skin contact on mother-preterm infant interaction through 18 months: randomized controlled trial. Int J Nurs Stud. 2009 Sep;46(9):1168-80. doi: 10.1016/j.ijnurstu.2009.03.005. Epub 2009 Apr 10. PMID 19361802